CLINICAL TRIAL: NCT04940208
Title: Chronic Pain in COVID-19 Patients Discharged From Intensive Care Unit - a Multicenter Observational Cohort Study
Brief Title: Chronic Pain in COVID-19 Patients Discharged From Intensive Care Unit
Status: Completed | Type: Observational
Sponsor: Mikhail Dziadzko, MD, PhD (Other)
Collaborators: Hôpital Raymond Poincaré (Other); Bicetre Hospital (Other)
Responsible Party: Sponsor-Investigator, Mikhail Dziadzko, MD, PhD, Attending Pain Physician, Hôpital de la Croix-Rousse
Organization: Hôpital de la Croix-Rousse (Other)
Other Study IDs: 2020-A02929-30
Record Dates: First submitted 2021-06-21; First posted 2021-06-25 (Actual); Last update posted 2022-02-02 (Actual); Status verified 2022-02

CONDITIONS: COVID-19 Pandemic; ICU; Pain, Chronic; Post Intensive Care Unit Syndrome; Neuropathic Pain
Keywords: SARS-COV2; Intensive care unit; critical illness survivors; chronic pain; COVID long; Neuropathic pain; Quantitative Sensory testing
MeSH Terms: conditions — COVID-19; Chronic Pain; Neuralgia; Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- post COVID-19 ICU survivors: Patients hospitalized to the ICU in the context of severe COVID-19 and discharged alive during the first French COVID-19 pandemic wave
  Interventions: Other: Pain and neuropsychological questionnaires; Diagnostic Test: Quantitative Sensory testing

INTERVENTIONS:
Other: Pain and neuropsychological questionnaires — Patient-reported outcomes, listed in the Secondary Outcome Measure Section
Diagnostic Test: Quantitative Sensory testing — Summation pain threshold test and Heat pain threshold skin test

SUMMARY:
More than six million French were affected by SARS-COV2 epidemic. About 20% of infected peoples were hospitalized, and about 5% were admitted to the intensive care units (ICU) for severe SARS-COV2 acute respiratory distress syndrome (ARDS) management.

A spectrum of neuropsychiatric sequelae, specific for the ICU exposure, was already described, including post-intensive care syndrome and persistent pain.

A growing body of evidence suggests the impact of SARS-COV2 exposure on the occurrence of neurological disorders and chronic pain syndrome development in COVID-19 patients.

Taking together, one can expect a large number of patients discharged from ICU after severe COVID-19 with high prevalence of persistent pain and psychological disorders. To date, no study has evaluated neither the incidence of persistant pains in ICU COVID-19 survivors, nor pain phenotypes.

The knowledge of such data is crucial in order to anticipate the management of such patients by specialized pain team, and to quantify the possible incurred burden of care.

Our study aims to evaluate the incidence of pain, pain localization and severity, associated pain-related psychological disorders, and to perform quantitative sensory testing in severe COVID-19 patients, admitted to the ICU for more than 48 hours and successfully discharged home during the first French pandemic wave.

ELIGIBILITY:
Inclusion Criteria:

* adults (>=18 y.o.)
* hospitalized in the ICU for at least 48 hours
* with SARS-Cov2 infection confirmed by Polymerase Chain Reaction (PCR)/serology and/or a suggestive chest Computed Tomography scan
* during the first wave of COVID 19 from March to December 2020 at three investigator sites (2 in Paris and 1 in Lyon)
* discharged alive from the ICU
* at least 6 months after discharge

Exclusion Criteria:

* patient refusal
* inability to communicate or to have in-person appointment
* death in the period from ICU discharge to the first phone call for interview

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: adult patients, infected with SARS COV2 and developed severe COVID, requiring hospitalisation to the ICU during the first French wave of COVID 19, with length of stay > 48 hours, survived and successfully discharged, and approached from 6th month post discharge.
Sampling Method: Non-Probability Sample
Enrollment: 143 (Actual)
Dates: Start 2021-01-11 (Actual); Primary Completion 2022-01-01 (Actual); Study Completion 2022-02-01 (Actual)

PRIMARY OUTCOMES:
Incidence of secondary chronic pain | starting 6 month after discharge
  Secondary chronic pain as defined by International Classification of Disease -11th revision (ICD-11).
  Chronic secondary pain is organized into the following six categories:
  1. Chronic cancer-related pain (ICD-11 code MG30.1)
  2. Chronic postsurgical or post-traumatic pain (ICD-11 code MG30.2)
  3. Chronic secondary musculoskeletal pain (ICD-11 code MG30.3)
  4. Chronic secondary visceral pain (ICD-11 code MG30.4)
  5. Chronic neuropathic pain (ICD-11 code MG30.5)
  6. Chronic secondary headache or orofacial pain (ICD-11 code MG30.6)
  Any pain detected in the population of interest and fitting in one of 6 categories will be accounted.

SECONDARY OUTCOMES:
Frequency of different secondary chronic pain classes | starting 6 month after discharge
  as defined by ICD-11 and the International Association for the Study of Pain (IASP)
  Chronic secondary pain is organized into the following six categories:
  1. Chronic cancer-related pain (ICD-11 code MG30.1)
  2. Chronic postsurgical or post-traumatic pain (ICD-11 code MG30.2)
  3. Chronic secondary musculoskeletal pain (ICD-11 code MG30.3)
  4. Chronic secondary visceral pain (ICD-11 code MG30.4)
  5. Chronic neuropathic pain (ICD-11 code MG30.5)
  6. Chronic secondary headache or orofacial pain (ICD-11 code MG30.6)
  For each category of detected pain the frequency will be reported.
Pain sensitivity level | starting 6 month after discharge
  Pain sensitivity level is tested with a Pain sensitivity questionnaire (PSQ). PSQ contains 17 items assessing pain with 11 level scoring from 0 (not at all painful) to 10 (most severe pain imaginable). Maximal summation score is 170, higher score mean worse outcome.
Pain localization | starting 6 month after discharge
  A Michigan Body Map will be used for pain localization inventory. A Michigan Body Map is a self-report measure to assess body areas where chronic pain is experienced.
The severity of pain and its impact on functioning | starting 6 month after discharge
  A Brief Pain Inventory (BPI) will be used to assess the severity of pain and its impact on functioning. The BPI pain scales defines pain as follows: Worst Pain Score: 1 - 4 = Mild Pain. Worst Pain Score: 5 - 6 = Moderate Pain. Worst Pain Score: 7 - 10 = Severe Pain. BPI Interference Items use 0 (less) to 10 (worth) scoring, the arithmetic mean of the interference items is used as a measure of pain interference, higher score mean worse outcome.
Neuropathic pain | starting 6 month after discharge
  A DN4 scale will be used to detect a neuropathic pain. The DN4 (which stands for Douleur Neuropathique 4) is a clinician-administered questionnaire consisting of 10 items. Seven items related to pain quality (i.e. sensory and pain descriptors) are based on an interview with the patient and 3 items based on the clinical examination. Each item has binary value (yes/no), maximal summation score is 10, and the threshold for neuropathic pain is 4.
Spiegel Sleep Quality Questionnaire | starting 6 month after discharge
  Spiegel Sleep Questionnaire is a self-rated questionnaire which assesses the current sleep quality and disturbances. It has six 5 point Likert-like items rated from worst to best value. The total summation score is 30, less score values indicates worth outcome. The threshold of bad sleep is less than 15, and the score 20 indicates a good sleep.
Posttraumatic Stress Disorder | starting 6 month after discharge
  Posttraumatic Stress Disorder Checklist Scale is a 20-item self-report measure that assesses the symptoms of Posttraumatic Stress Disorder. Respondents rate each item from 0 ("not at all") to 4 ("extremely") to indicate the degree to which they have been bothered by that particular symptom over the past month.
  A total symptom severity score is obtained by summing the scores for each of the 20 items. The score superior of 31 is indicative of probable Posttraumatic Stress Disorder.
Anxiety and Depression | starting 6 month after discharge
  Hospital Anxiety Depression scale will be used, it measures anxiety and depression in a general medical population of patients. The questionnaire comprises seven questions for anxiety and seven questions for depression. Greater score values indicates worth outcome.
  For both scales, scores of less than 7 indicate non-cases; 8-10 - mild depression or anxiety; 11-14 - moderate depression or anxiety; and 15-21 - severe depression or anxiety.
Pain Catastrophizing Level | starting 6 month after discharge
  Pain Catastrophizing Scale quantifies an individual's pain experience. It has 13 items rated on 5-point Likert-like scales (0 - not at all to 4 - all the time). A total score is yielded (ranging from 0-52), the threshold above 30 is considered clinically relevant. Higher score indicates higher level of catastrophizing and bad outcome.
Perceived Stress Level | starting 6 month after discharge
  Perceived Stress Scale (PSS-10) is a self stress assessment instrument. It has 10 items rated on 5-point Likert-like scales (0 - never to 4 - very often). Individual scores on the PSS-10 can range from 0 to 40 with higher scores indicating higher perceived stress.
Summation pain threshold | starting 6 month after discharge
  Mechanical temporal summation will be evoked using methodology described by Weissman-Fogel, 2008, by Von Frey Filaments, using a 180-gr filament that will be applied to the volar aspect of the dominant forearm. Patients will be exposed to a single stimulus and will be asked to rate the level of pinprick pain intensity using 11 items numeric pain scale. This pain score serve as an index for mechanical suprathreshold pain. Subsequently, 1 Hz repetitive stimuli will be applied within an area of 1 cm in diameter, using the same filament, and subjects will be asked to rate the pain intensity of the last stimulus. The magnitude of mechanical temporal summation will be calculated as the difference between the last and the first pain scores. Higher values indicates worth outcome.
Heat pain threshold | starting 6 month after discharge
  A heat pain threshold will be realized using Thermal Stimulator for Sensory testing (SOMEDIC(R)). A thermode (heating stick) of 7 square centimeters will be applied to the volar aspect of the dominant forearm. Patients will be exposed to 3 repetitive gradual increase in temperature from 32° to 52°C. The skin contact will be withdrawn if an individual is not able to tolerate such stimulation, and the temperature threshold of tolerance will be noted. The final reading will be the median of three measurements, higher values indicate better tolerance.

CONTACTS AND LOCATIONS:
Locations (3):
- France (3):
  - Hôpital Raymond Poincare - AP-HP, Garches, Hauts-de-Seine
  - Hôpital Bicêtre AP-HP, Le Kremlin-Bicêtre
  - Hopital de la Croix Rousse - Hospices Civils de Lyon, Lyon

IPD SHARING:
Plan to Share IPD: No
individual participant data are the property of investigator's centers and will not be shared

REFERENCES:
- [Background] Carfi A, Bernabei R, Landi F; Gemelli Against COVID-19 Post-Acute Care Study Group. Persistent Symptoms in Patients After Acute COVID-19. JAMA. 2020 Aug 11;324(6):603-605. doi: 10.1001/jama.2020.12603. PMID 32644129
- [Background] Needham EJ, Chou SH, Coles AJ, Menon DK. Neurological Implications of COVID-19 Infections. Neurocrit Care. 2020 Jun;32(3):667-671. doi: 10.1007/s12028-020-00978-4. PMID 32346843
- [Background] Asadi-Pooya AA, Simani L. Central nervous system manifestations of COVID-19: A systematic review. J Neurol Sci. 2020 Jun 15;413:116832. doi: 10.1016/j.jns.2020.116832. Epub 2020 Apr 11. PMID 32299017
- [Background] Lee AM, Wong JG, McAlonan GM, Cheung V, Cheung C, Sham PC, Chu CM, Wong PC, Tsang KW, Chua SE. Stress and psychological distress among SARS survivors 1 year after the outbreak. Can J Psychiatry. 2007 Apr;52(4):233-40. doi: 10.1177/070674370705200405. PMID 17500304
- [Derived] Martinez V, Dziadzko M, Tamayo J, Schitter S, Guichard L, Richeux F, Roggerone S, Branche P, Schlaefflin L, Nacto Y, Antunes T, Negre I, Annane D, Aubrun F. Chronic pain characteristics in COVID-19 survivors after an ICU stay. A cross-sectional study. Anaesth Crit Care Pain Med. 2023 Dec;42(6):101267. doi: 10.1016/j.accpm.2023.101267. Epub 2023 Jun 24. PMID 37356618